CLINICAL TRIAL: NCT05070104
Title: Phase I Study of the First-In-Class Agent CPI-613 (Devimistat) in Combination With Modified FOLFIRINOX Plus Bevacizumab in Patients With Metastatic Colorectal Cancer
Brief Title: CPI-613 (Devimistat) in Combination With Modified FOLFIRINOX Plus Bevacizumab in Patients With Metastatic Colorectal Cancer
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: no funding
Sponsor: Cornerstone Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACHIEVE613
Record Dates: First submitted 2021-09-17; First posted 2021-10-06 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: C04.588.274.476.411.307
MeSH Terms: interventions — devimistat; Bevacizumab

STUDY DESIGN:
Intervention Model Description: Single group, Open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental): CPI-613 mFFX Bevacizumab
  Interventions: Drug: CPI-613; Drug: modified FFX; Drug: Bevacizumab

INTERVENTIONS:
Drug: CPI-613 — 250-1000mg/m2 -14 day cycle
  Other Names: Devimistat
Drug: modified FFX — Irinotecan: 150mg/m2 IV over 90 min-14 day cycle Leucovorin: 400mg/m2 IV over 2hrs with Irinotecan-14 day cycle Oxaliplatin: 85mg/m2 IV over 2hrs-14 day cycle 5FU: 2400mg/m2 IV over 46-48 hrs-14 day cycle
Drug: Bevacizumab — 5mg/kg IV

SUMMARY:
Pre-clinical in vitro and in vivo data as well as early phase 1 clinical trials have shown that both hematologic and solid tumor cells are susceptible to single-agent cytotoxicity by CPI-613 (devimistat), consistent with its selective target of the altered form of mitochondrial energy metabolism in tumor cells, causing changes in mitochondrial enzyme activities and redox status, which lead to apoptosis, necrosis, and autophagy of tumor cells leading to the death of cancer cells. It is our hypothesis that CPI-613 (devimistat) will enhance the efficacy of mFOLFIRINOX plus Bevacizumab when given as a combination treatment. The study will follow a standard 3+3 design. Cohorts of three to six patients will be treated at each dose level until the MTD is defined.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent in accordance with federal, local, and institutional guidelines
2. Patients must have histologically/pathologically confirmed colorectal adenocarcinoma with measurable disease by RECIST 1.1 criteria
3. Patients must have had no prior chemotherapy for metastatic disease with fluoropyrimidine based chemotherapy with oxaliplatin or irinotecan
4. Patients with prior adjuvant chemotherapy are allowed, as long as a minimum of 6 months have passed between the completion of adjuvant therapy and the start of the study medication
5. Age >18 years
6. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
7. Radiographic evidence of metastatic disease
8. At the time of study entry:

   absolute neutrophil count must be ≥ 1000/mm3, hemoglobin ≥ 9 gm/dL, and platelet count ≥ 100,000/mm3 There must be evidence of adequate hepatic and renal function. Bilirubin must be ≤ 1.5 x upper limit of normal (ULN) for the lab unless the patient has a chronic grade 1 bilirubin elevation due to Gilbert's disease or similar syndrome due to slow conjugation of bilirubin Alkaline phosphatase must be ≤ 3 x ULN for the lab AST and ALT must be ≤ 5 x ULN for the lab Serum creatinine ≤ 1.5 x ULN for the lab Note: For patients with liver metastases, non-fasting bilirubin 1.5 x ULN to 3 x ULN of the institution's normal range are acceptable.
9. Both male and female patients with childbearing potential must agree to use adequatecontraception throughout the study and for 9 months after last dose of mFOLFIRINOX, bevacizumab or CPI-613 (devimistat)
10. Patients without liver metastasis are eligible if they have ALT and AST ≤ 3.0 x ULN

Exclusion Criteria:

1. Diagnosis of anal or small bowel carcinoma
2. Colorectal cancer other than adenocarcinoma, e.g., sarcoma, lymphoma, carcinoid
3. Patients with tumors that are MSI-high/dMMR
4. Receipt of live attenuated vaccination within 30 days prior to study entry or within 30 days ofreceiving study therapy
5. Active infection or chronic infection requiring systemic therapy
6. Known history of human immunodeficiency virus (HIV) or acquired immunodeficiencyrelated (AIDS) illnesses with CD4 count < 250 cells/mm3
7. Any of the following cardiac conditions:

   Documented NYHA Class III or IV congestive heart failure, Myocardial infarction within 6 months prior to study entry, Unstable angina within 6 months prior to study entry, Symptomatic arrhythmia
8. Other malignancies unless the patient is considered to be disease-free and has completed therapy for the malignancy ≥ 12 months prior to study entry.

   Patients with the following cancers are eligible if diagnosed and treated within the past 12 months: carcinoma in situ of the cervix, and basal cell and squamous cell carcinoma of the skin
9. Psychiatric or addictive disorders or other conditions that in the opinion of the investigator would preclude the patient from meeting the study requirements or interfere with interpretation of study results
10. Any other chronic or clinically significant medical condition that in the opinion of investigator would jeopardize the safety or rights of the volunteer. Including, but not limited to: diabetes mellitus type I, chronic hepatitis; OR clinically significant forms of drug oralcohol abuse, asthma, autoimmune disease, psychiatric disorders, heart disease, or cancer. Patients must have neuropathy grade 1 or less
11. Pregnancy or lactation at the time of study entry
12. Use of any investigational agent within 4 weeks prior to the first dose study therapy
13. Patients with the following conditions:

    Uncontrolled hypertension (defined as systolic blood pressure ≥ 150 mm Hg and diastolic blood pressure ≥ 100 mm Hg) Bleeding diatheses or hemorrhage within 6 months prior of study enrollment Gastrointestinal perforation or fistulas History of thromboembolic events Reversible Posterior Leukoencephalopathy Syndrome (RPLS), Proteinuria > 1gr/24 hours
14. Patients with current serious, non-healing wound, ulcer and baseline peripheral neuropathy of grade 2 or greater, hypersensitivity reaction to 5-FU, oxaliplatin or other platinum-based drugs, or irinotecan if it was previously administered in the adjuvant setting

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-03-30 (Estimated); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability | 3-6 months
  Number of patients with Dose-limiting toxicities (DLT) will be assessed in order to be able to establish safety and tolerability for the combination of CPI-613, mFFX with bevacizumab therapy. Using the descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 for adverse event reporting (Grade 1 (Mild) - 5 (Death) as well as expectedness (unexpected/expected) and attribution (definitely related to study treatment to unrelated to study treatment).
Safety and tolerability | 3-6 months
  Dose-limiting toxicities assessed in order to be able to establish safety and tolerability for the combination of CPI-613, mFFX with bevacizumab therapy. Using the descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 for adverse event reporting (Grade 1 (Mild) - 5 (Death) as well as expectedness (unexpected/expected) and attribution (definitely related to study treatment to unrelated to study treatment).
Recommended Phase 2 Dose | 3-6 months
  Determine recommended phase 2 dose (RP2D) of CPI-613 (devimistat) (MTD) in combination with mFOLFIRINOX plus bevacizumab

SECONDARY OUTCOMES:
Objective Response Rate | 3-12 months
  It is defined as the proportion of patients who achieve complete response or partial response during or following study treatment
Overall Survival | 3-12 months
  Defines as the time from enrollment to the date of death due to any cause.

IPD SHARING:
Plan to Share IPD: Undecided